CLINICAL TRIAL: NCT06623786
Title: Cancer Patient Remote Monitoring for Timely Communication Study
Acronym: CONNECT
Status: Not yet recruiting | Type: Observational
Sponsor: Asklepios proresearch (Industry)
Collaborators: Q1.6 B.V. (Unknown); Medical University of Vienna (Other)
Responsible Party: Sponsor
Other Study IDs: The CONNECT Study
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-08

CONDITIONS: NSCLC Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Double immune checkpoint inhibitor: * Histologically or cytologically confirmed stage IV NSCLC without EGFR sensitizing mutations or ALK translocations OR
  * Histologically or cytologically confirmed advanced, malignant pleural mesothelioma
  * Eligible for double immune checkpoint inhibition with an anti PD1/L1 inhibitor and a CTLA-4 inhibitor with or without chemotherapy according to current guidelines and SmPC
- Immunotherapy with PD1/L1 inhibitor: * Histologically or cytologically confirmed stage IV NSCLC without EGFR sensitizing mutations or ALK translocations
  * Eligible for treatment with an anti-PD-1/L1 inhibitor with or without chemotherapy according to current guidelines and SmPCs

SUMMARY:
The study is designed as a prospective, single-arm observational, mixed-method study. Patients with stage IV NSCLC or inoperable mesothelioma will be included and will be treated with immunotherapy according to current guidelines and standard of care. Patients may receive either a PD1/L1 inhibitor monotherapy or, if indicated, together with a CTLA4 inhibitor. Immunotherapy may be administered alone or together with chemotherapy as per site standard/physician's choice. Patients will be given access to a mobile app. Patients will receive daily questions via the app to assess immune-related adverse events between clinic visits and their well-being.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age > 18 years at the time of study entry
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Life expectancy > 6 months
* Patient is able and willing to use smart phone and a wearable device/technology/sensor

Exclusion Criteria:

* Previous systemic treatment for metastatic or locally advanced disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort 1: Double immune checkpoint inhibition
  * Histologically or cytologically confirmed stage IV NSCLC without EGFR sensitizing mutations or ALK translocations OR
  * Histologically or cytologically confirmed advanced, malignant pleural mesothelioma
  * Eligible for double immune checkpoint inhibition with an anti PD1/L1 inhibitor and a CTLA-4 inhibitor with or without chemotherapy according to current guidelines and SmPCs
  Cohort 2: Immunotherapy with PD1/L1 inhibitor:
  * Histologically or cytologically confirmed stage IV NSCLC without EGFR sensitizing mutations or ALK translocations
  * Eligible for treatment with an anti-PD-1/L1 inhibitor with or without chemotherapy according to current guidelines and SmPCs
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
adherence to use the remote monitoring app | 6 months
  To measure the adherence to use the remote monitoring app, assessed as percentage of answered questions related to the total number of questions sent to the patients via Q1.6 app

IPD SHARING:
Plan to Share IPD: No